CLINICAL TRIAL: NCT01055639
Title: Telehealth Therapy for Chronic Pain
Brief Title: Telehealth Therapy for Chronic Pain: Comparison of In-person vs. Video-administered ACT for Pain
Acronym: TTCP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F6891-R; 091019 (Other Grant/Funding Number: GRANT00557035)
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Acceptance and Commitment Therapy (ACT)
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In-person ACT (Active Comparator): 8 individual in-person sessions of Acceptance and Commitment Therapy (ACT). ACT is a psychotherapy intervention comprised of meditation, goal-setting, and behavior change.
  Interventions: Behavioral: In-Person ACT
- Telehealth ACT (Experimental): 8 individual telehealth sessions of Acceptance and Commitment Therapy (ACT). Sessions were delivered via videoconferencing system. ACT is a psychotherapy intervention comprised of meditation, goal-setting, and behavior change.
  Interventions: Behavioral: Telehealth ACT

INTERVENTIONS:
Behavioral: In-Person ACT — 8 individual in-person sessions of Acceptance and Commitment Therapy (ACT): includes mindfulness, values, and committed action
  Arms: In-person ACT
Behavioral: Telehealth ACT — 8 individual telehealth sessions of Acceptance and Commitment Therapy (ACT): includes mindfulness, values, and committed action
  Arms: Telehealth ACT

SUMMARY:
The purpose of the study is to test a brief, individual psychosocial in-person or telehealth intervention to reduce interference of pain with daily life, emotional distress, and pain intensity, and improve quality of life and physical activity levels in individuals with chronic pain.

DETAILED DESCRIPTION:
Chronic pain affects at least 15% of the veteran population and represents a high priority for the VA. In addition to primary pain conditions, chronic pain is a common secondary condition resulting from battlefield injuries, traumatic accidents, and congenital and acquired disorders. Unlike most forms of acute pain, treatment options available for patients suffering from chronic pain frequently offer only short-term or partial relief from symptoms. The focus of rehabilitative intervention thus becomes the reduction of disability and emotional distress and improvement in quality of life and activity levels.

Chronic pain rehabilitation has evolved from a primarily one dimensional, medically oriented approach to a multidisciplinary approach that incorporates a biopsychosocial formulation to pain management with physiological, cognitive, behavioral, and emotional components. This conceptualization of pain recognizes that multiple intervention modalities, including psychosocial approaches, are required when providing treatment to chronic pain patients.

A relatively new psychosocial approach to chronic pain management and rehabilitation involves acceptance of pain-related experiences. The Acceptance and Commitment Therapy (ACT) model is based on the theory that attempts to escape, avoid, or control negative experiences that cannot be changed, such as chronic pain, may paradoxically contribute to the increased experience of them. Instead of seeking to control the negative experience, ACT teaches individuals to use mindfulness strategies to enlarge the scope of experience beyond pain and to engage in behaviors that are consistent with personal values and goals when total elimination of pain or other negative experiences is not possible. Empirical support for acceptance-based approaches to chronic pain management is growing. Data from one of the first comparisons of ACT to a well-established psychosocial intervention, Cognitive-Behavioral Therapy (CBT), performed at the VA San Diego Healthcare System (VASDHS) by the PI, suggests that ACT may be superior to CBT as an adjunctive treatment for chronic pain.

The proposed study assembles a multidisciplinary team with extensive experience in chronic pain interventions research to evaluate the benefits of a brief, individual psychosocial in-person or telehealth intervention which could be easily integrated into multidisciplinary pain rehabilitation programs throughout the VA system to reduce disability in veterans with chronic pain secondary to other conditions. Specifically, we propose to examine the effects of a promising new chronic pain intervention based on ACT principles on the primary outcome of pain interference and secondary outcomes of emotional distress, quality of life, physical activity, pain intensity, and treatment satisfaction among 196 veterans with chronic benign pain as a secondary condition. The participants are randomized to between-subjects design where in-person ACT intervention will be compared with telehealth ACT intervention. Outcomes include an objective measure of physical activity, actigraphy, as well as self-reported measures and will be evaluated at baseline, 4 weeks, 8 weeks (end of treatment), 3-month follow-up and at a 6-month follow-up period to investigate maintenance of gains. Telehealth sessions are conducted using secure video-conferencing equipment at the most convenient clinic for the participant. Thus, the proposed project has the potential to enhance the current VA standard of care as well as to add to the scientific literature on psychological models and rehabilitation of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-terminal pain condition;
* Pain severity and interference rated > 4/10; and
* Pain most days (> 3/week) for at least 6 months.

Exclusion Criteria:

* Current participation in group psychotherapy for pain or any type of individual psychotherapy;
* Previous treatment with ACT;
* Active suicide ideation or history of suicide attempt within 5 years;
* Serious or unstable medical or psychiatric illness or psychosocial instability that could compromise study participation; and
* The following DSM-IV diagnoses or active problems within the past 6 months noted in the patient's Computerized Patient Record System (CPRS) medical record or diagnosed during a structured psychiatric interview:

  * schizophrenia;
  * other psychotic disorder;
  * bipolar disorder;
  * organic mental disorder;
  * borderline or antisocial personality disorder; or
  * alcohol or substance abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Wetherell, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Herbert MS, Afari N, Liu L, Heppner P, Rutledge T, Williams K, Eraly S, VanBuskirk K, Nguyen C, Bondi M, Atkinson JH, Golshan S, Wetherell JL. Telehealth Versus In-Person Acceptance and Commitment Therapy for Chronic Pain: A Randomized Noninferiority Trial. J Pain. 2017 Feb;18(2):200-211. doi: 10.1016/j.jpain.2016.10.014. Epub 2016 Nov 9. PMID 27838498

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In-person ACT | Telehealth ACT
Started | 66 | 60
Completed | 45 | 31
Not Completed | 21 | 29
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 8 | 11
Not completed — Protocol Violation | 5 | 5
Not completed — Withdrawal by Subject | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-person ACT | Telehealth ACT | Total
Number analyzed (Participants) | 66 | 60 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 54 | 109
  >=65 years | 11 | 6 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 55 | 50 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 19
  Not Hispanic or Latino | 55 | 52 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 19 | 16 | 35
  White | 38 | 33 | 71
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory-interference Subscale
Description: The primary outcome measure for the proposed study is the Brief Pain Inventory Short Form Interference subscale (BPI; Cleeland & Ryan, 1994). This 7-item scale, recommended by the IMMPACT group as a measure of functioning (Dworkin et al., 2005), measures the degree to which pain interferes with various aspects of life, including mobility, social activities, and mood. Scores range from 0 (least interference due to pain) to 10 (most interference due to pain).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 5.3 (2.4) | 5.8 (2.3)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

2. Secondary Outcome: Brief Pain Inventory-severity Subscale
Description: The Brief Pain Inventory Short Form (BPI; Cleeland & Ryan, 1994) includes a 4-item pain severity subscale measuring the level of pain over the past week on average, at its worst, at its least, and currently. This measure is recommended by the IMMPACT group as a pain assessment tool (Dworkin et al., 2005). Scores range from 0 (least pain severity) to 10 (most pain severity).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 5.2 (1.7) | 5.7 (1.5)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

3. Secondary Outcome: West Haven-Yale Multidimensional Pain Inventory - Activity Subscales
Description: The West Haven-Yale Multidimensional Pain Inventory (MPI; Kerns et al., 1985) contains 52 items forming 12 subscales. For this study, we used four subscales assessing various types of activities. Household Chores (5 items); Outdoor Work (5 items); Activities Away From Home (4 items); and Social Activities (4 items). The MPI has been used extensively in outcome research with heterogeneous samples of chronic pain patients, including veterans, and has demonstrated sensitivity to treatment change (Altmaier et al., 1992; Mikail et al., 1993). Individual items are rated on a 7-point Likert scale from 0-6, and subscales are scored by averaging items together. Therefore, the score for Part III, General Activity, is composed of an average of the 18 items in the Household Chores (5 items); Outdoor Work (5 items); Activities Away From Home (4 items); and Social Activities (4 items) subscales. The final score ranges from 0 (lowest level of activity) to 6 (highest level of activity).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 2.4 (1.0) | 2.2 (0.9)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.88, t-test, 2 sided

4. Secondary Outcome: SF-12 MCS
Description: 6-item self-report measure of mental health-related quality of life. Subscale of the Medical Outcomes Study 12-Item Short Form Health Survey (SF-12; Ware et al., 1994). This measure is widely used with populations with chronic disease. The Physical and Mental Component Summary scores correlate .91 and .92 with the corresponding scores derived from the SF-36, and 2-week test-retest reliability correlations were .89 and .76 (Ware et al., 1994). The Short Form Health Survey is recommended by the IMMPACT group (Dworkin et al., 2005). Scores range from 0 (lowest functioning) to 100 (highest functioning).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 41.5 (12.9) | 41.6 (12.8)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.48, t-test, 2 sided

5. Secondary Outcome: SF-12 PCS
Description: Physical health-related quality of life will be measured using the Physical Component Summary score of the Medical Outcomes Study 12-Item Short Form Health Survey (SF-12; Ware et al., 1994). This measure is widely used with populations with chronic disease. The Physical and Mental Component Summary scores correlate .91 and .92 with the corresponding scores derived from the SF-36, and 2-week test-retest reliability correlations were .89 and .76 (Ware et al., 1994). The Short Form Health Survey is recommended by the IMMPACT group (Dworkin et al., 2005). Scores range from 0 (lowest functioning) to 100 (highest functioning).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 32.6 (9.3) | 30.9 (7.2)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.87, t-test, 2 sided

6. Secondary Outcome: Patient Health Questionnaire-9
Description: The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. The tool rates the frequency of the symptoms which factors into the scoring severity index. Scores range from 0 (lowest level of depressive symptoms) to 27 (highest level of depressive symptoms).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 9.6 (6.3) | 10.2 (6.1)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.29, t-test, 2 sided

7. Secondary Outcome: Pain Anxiety Symptom Scale - 20
Description: Anxiety will be assessed with the 20-item Pain Anxiety Symptoms Scale-Short Form (PASS-20; McCracken & Dhingra, 2002). Pain anxiety captures fears patients associate with their symptoms, which are typically associated with the belief that their pain signals harm. High levels of pain anxiety compromise patient's activity levels, participation in rehabilitation, and performance on functional tests. The instrument is a valid and reliable measure of anxiety symptoms in pain populations (McCracken et al., 1996; Roelofs et al., 2004). The PASS-20 items are scored on a 6-point Likert scale and assess cognitive, escape/avoidance, fear, and physiological anxiety dimensions. Internal consistency is high and correlation between the short and long form is excellent (alpha=.81; r=.97). This measure has been recommended by the VA and demonstrated sensitivity to treatment in the pilot sample (National VA Pain Outcomes Working Group, 2003). Scores range from 0 (least anxiety) to 100 (most anxiety).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 39.8 (24.4) | 43.5 (23.0)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.19, t-test, 2 sided

8. Secondary Outcome: PTSD Checklist
Description: The 17-item PTSD Checklist (Weathers et al., 1994) will be used to assess PTSD symptoms. In combat veterans, this questionnaire has high test-retest reliability (0.96) and validity as indicated by a kappa of 0.64 for diagnosis of PTSD using the SCID (Weathers et al., 1993). Scores range from 17 (low PTSD) to 85 (high PTSD).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 42.7 (17.2) | 42.5 (17.3)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 0.53, t-test, 2 sided

9. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: The 19-item Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989) is the most commonly used measure of self-rated sleep quality, with good reliability (alpha = .83, test-retest = .85) and validity (kappa = 0.75) for distinguishing good and poor sleepers. A survey recently conducted by the IMMPACT group indicated that sleep is one of the domains most important to patients with chronic pain (Turk et al., 2008), and the PSQI is the scale most frequently used to evaluate sleep quality in studies of chronic pain patients (Cole et al., 2007). Scores range from 0 (good sleep) to 42 (poor sleep).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-person ACT | Telehealth ACT
Number analyzed (Participants) | 66 | 60
units on a scale | 11.8 (4.6) | 11.8 (4.1)
Statistical Analysis 1: Comparison: In-person ACT vs Telehealth ACT; Test type: Superiority or Other; p = 1.00, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks (duration of intervention)
Arm/Group | In-person ACT | Telehealth ACT
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/60
Other Adverse Events (participants affected / at risk) | 0/66 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-person ACT (N=66) | Telehealth ACT (N=60)
hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — One person in the telepain group experienced increased anxiety and was hospitalized overnight

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No